CLINICAL TRIAL: NCT05521919
Title: Effects of Acute Stress Exposure on Plasma Beta-amyloid Levels
Brief Title: Acute Plasma Abeta Responses to Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Washington University School of Medicine (Other); Keck School of Medicine of USC (Other)
Responsible Party: Principal Investigator, Mara Mather, Professor of Gerontology, Psychology, and Biomedical Engineering, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP-22-00404
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Stress Reaction; Stress Physiology
Keywords: Stress Reaction; Stress; Amyloid-Beta
MeSH Terms: conditions — Fractures, Stress; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Participants will complete one session of each condition: stress and no-stress. Participants will be randomly assigned to one of the two conditions for their first session. Participants will then be randomly assigned to the remaining condition for the second session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress (sympathetic nervous system activation) (Experimental): Stress will be induced using the socially evaluated cold pressor test.
  Participants will complete three rounds of the socially evaluated cold pressor test.
  The socially evaluated cold pressor test involves submerging one hand in ice-cold water for 3 minutes while participants' reactions are filmed on camera.
  Interventions: Behavioral: Sympathetic Nervous System Activation
- No-stress (Sham Comparator): Participants will hold a hand in room temperature water for 3 minutes.
  Interventions: Behavioral: No-stress

INTERVENTIONS:
Behavioral: Sympathetic Nervous System Activation — Participants will complete a task that increases sympathetic nervous system activation.
  Arms: Stress (sympathetic nervous system activation)
Behavioral: No-stress — Participants will complete a task that will not affect their sympathetic nervous system activity.
  Arms: No-stress

SUMMARY:
Research has shown that activation of the sympathetic nervous system for extended periods or during certain times in life can increase the risk for Alzheimer's disease. Some research in animal models show that acute activation of the sympathetic nervous system through stress exposure can increase certain Alzheimer's disease-related biomarkers, such as amyloid-beta, within hours of exposure. However, how acute sympathetic nervous system activation via stress exposure affects amyloid-beta levels in humans has yet to be examined.

In this study, the investigators will examine whether brief increases in sympathetic activation result in immediate changes in plasma amyloid-beta levels in the five hours after exposure.

DETAILED DESCRIPTION:
Aim 1: determine whether acute exposure to stress (increasing sympathetic nervous system activation) increases plasma amyloid-beta-40 and amyloid-beta-42 in the five hours following exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult weighing at least 110 pounds
* No chronic conditions or illness
* Taking no medications or drugs that might alter the stress response (e.g., corticosteroids, beta-blockers, and others)
* Not using any hormone-containing medication (e.g., hormonal contraceptives, hormone replacement, etc.)
* No contraindications for cold pressor test exposure (high blood pressure, heart disease, dysrhythmia, peripheral vascular disease, any other cardiovascular disorder, diabetes, vasculitis, lupus, tingling or numbness in the hands and/or feet, cryoglobulinemia, and Reynaud's phenomenon)
* No history of fainting during blood draws
* No phobia of having their blood drawn
* No general history of fainting or seizures
* Not currently diagnosed with a mood disorder (e.g., major depressive disorder)
* Not pregnant in the past 12 months
* Not lactating in the past 12 months
* Not trying to become pregnant if premenopausal
* Experienced natural menopause if postmenopausal
* Be non-smokers
* Be fluent in English

Exclusion Criteria:

- Unwilling to be filmed during the stress task OR unwilling to sign the waiver allowing their filmed responses to be used in scientific presentations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Plasma amyloid-beta-40 | 9.5 hours
  Changes in levels of amyloid-beta-40 in blood from before to after acute intervention (stress/no-stress).
Plasma amyloid-beta-42 | 9.5 hours
  Changes in levels of amyloid-beta-42 in blood from before to after acute intervention (stress/no-stress).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data (values of outcome measures and associated experimental conditions) will be shared publicly on Open Science Framework.
Time Frame: Data will be made available by publication of the paper reporting on the results.
Access Criteria: Publicly available.